CLINICAL TRIAL: NCT00743691
Title: Impact of Strengthened Health Extension Program and Community Based Treatment of Neonatal Infections on Neonatal Mortality in Oromia and South Nation and Nationalities & People Region(SNNPR), Ethiopia
Brief Title: Impact Study of Community Based Treatment of Neonatal Infection by Health Extension Workers on Neonatal Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Save the Children (Other)
Collaborators: John Snow, Inc. (Industry); University of London (Other); UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: SNL 50124
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Neonatal Infections
Keywords: Ethiopia; Community; Community based; Health extension Worker; Health Extension Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1 (No Intervention): Make a diagnosis of Neonatal infections and refer patients according to IMNCI guideline
- 2 (Active Comparator): Health extension Workers will Make a diagnosis of Neonatal infections and treat with antibiotics when referal is not possible
  Interventions: Other: Community Based

INTERVENTIONS:
Other: Community Based — In Arm 2 health extension workers will make a diagnosis of Neonatal infection and treat with antibiotics
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether community based management of infections with antibiotics administered by health extension workers reduce all cause mortality in neonates after the first day of life compared to current MOH IMNCI model of referral to hospital

DETAILED DESCRIPTION:
Although 44% of neonatal deaths in Ethiopia are due to infection, access to treatment for neonatal infections is very low for most families. Even though the newly adapted Integrated Management of Newborn and Childhood Illness (IMNCI) package includes assessment of newborns, if a baby has any danger signs that may be suggestive of infection and is taken to health posts, the baby is to be referred to hospital for treatment. Given that only about 5% of neonatal deaths occur in hospitals and the distance to hospital is often far and the costs prohibitive, very few babies are likely to receive essential lifesaving antibiotics. Evidence from India, Bangladesh, and Nepal demonstrates that community health workers can effectively manage neonatal infections at home. However it is not known whether and community-based management of neonatal infections is effective, feasible and acceptable in the Ethiopian context. Local evidence regarding lives saved and cost is required in order to inform health policy and programming regarding community-based treatment of neonatal infections.

ELIGIBILITY:
Inclusion Criteria:

* Participants who give consent to be treated at Health Post by Health extension worker

Exclusion Criteria:

* If Newborn is Critically sick

Ages: 1 Minute to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19476 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All cause Neonatal Mortality | 2 years

SECONDARY OUTCOMES:
Additional cost for community based neonatal infection management | 2 years
Adding identification and treatment of newborns and children to the package of services provided by HEWs/CHPs will not adversely affect the coverage of other services currently provided. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T. Tesema, MD,Ped, Principal Investigator — Save the Children; Brian E. Mulligan, BSc, MPH, Principal Investigator — John Snow, Inc.; Tedbab D. HaileGebreil, MD, Ped, Principal Investigator — Save the Children/USA Ethiopia country office; Simon Ni Cousens, professor, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Sidama, East shoa and West arsi Zones, Ādama, Sidama Region, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed S, Sobhan F, Islam A, Barkat-e-Khuda. Neonatal morbidity and care-seeking behaviour in rural Bangladesh. J Trop Pediatr. 2001 Apr;47(2):98-105. doi: 10.1093/tropej/47.2.98. PMID 11336143
- [Background] Baqui AH et al. Early Findings from a Cluster-randomized Community-based Newborn Health Intervention Trial in Sylhet, Bangladesh. 8th Commonwealth Congress on Diarrhoea and Malnutrition (CAPGAN), 2006
- [Background] Bang AT, Bang RA, Baitule SB, Reddy MH, Deshmukh MD. Effect of home-based neonatal care and management of sepsis on neonatal mortality: field trial in rural India. Lancet. 1999 Dec 4;354(9194):1955-61. doi: 10.1016/S0140-6736(99)03046-9. PMID 10622298
- [Background] Bhutta ZA, Darmstadt GL, Hasan BS, Haws RA. Community-based interventions for improving perinatal and neonatal health outcomes in developing countries: a review of the evidence. Pediatrics. 2005 Feb;115(2 Suppl):519-617. doi: 10.1542/peds.2004-1441. PMID 15866863
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Lawn JE and Kerber K (eds) .Opportunities for Africa's Newborns: Practical data, policy and programmatic support for newborn care in Africa. The Partnership for Maternal, Newborn & Child Health (PMNCH), Cape Town 2006. ISBN-13: 978-0-620-37695-2.
- [Background] Lawn JE, Wilczynska-Ketende K, Cousens SN. Estimating the causes of 4 million neonatal deaths in the year 2000. Int J Epidemiol. 2006 Jun;35(3):706-18. doi: 10.1093/ije/dyl043. Epub 2006 Mar 23. PMID 16556647
- [Background] FMOHa. Health Sector Development Programme -III Document. Federal Ministry of Health, Addis Ababa, Ethiopia, November 2005.
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Derived] Degefie Hailegebriel T, Mulligan B, Cousens S, Mathewos B, Wall S, Bekele A, Russell J, Sitrin D, Tensou B, Lawn J, de Graft Johnson J, Legesse H, Hailu S, Nigussie A, Worku B, Baqui A. Effect on Neonatal Mortality of Newborn Infection Management at Health Posts When Referral Is Not Possible: A Cluster-Randomized Trial in Rural Ethiopia. Glob Health Sci Pract. 2017 Jun 27;5(2):202-216. doi: 10.9745/GHSP-D-16-00312. Print 2017 Jun 27. PMID 28611102
- See also: Official website for Save the Children — http://www.savethechildren.org